CLINICAL TRIAL: NCT01125800
Title: A Phase I/II Study of LDE225 in Pediatric Patients With Recurrent or Refractory Medulloblastoma or Other Tumors Potentially Dependent on the Hedgehog-signaling Pathway and Adult Patients With Recurrent or Refractory Medulloblastoma
Brief Title: A Phase I Dose Finding and Safety Study of Oral LDE225 in Children and a Phase II Portion to Assess Preliminary Efficacy in Recurrent or Refractory MB
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLDE225X2104; 2010-019348-37 (EudraCT Number)
Record Dates: First submitted 2010-05-12; First posted 2010-05-18 (Estimated); Results first posted 2016-03-02 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2016-02

CONDITIONS: Medulloblastoma; Rhabdomyosarcoma; Neuroblastoma; Hepatoblastoma; Glioma; Astrocytoma
Keywords: Recurrent,; refractory,; medulloblastoma,; rhabdomyosarcoma,; neuroblastoma,; hepatoblastoma,; astrocytoma,; children,; pediatric,; hedgehog pathway inhibitor, adult
MeSH Terms: conditions — Medulloblastoma; Rhabdomyosarcoma; Neuroblastoma; Hepatoblastoma; Glioma; Astrocytoma; Recurrence | interventions — sonidegib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- LDE225 233mg/m2 daily dose (Experimental): Pediatric dose.
  Interventions: Drug: LDE225
- LDE225 372mg/m2 daily dose (Experimental): Pediatric dose.
  Interventions: Drug: LDE225
- LDE225 425 mg/m2 daily dose (Experimental): Pediatric dose.
  Interventions: Drug: LDE225
- LDE225 680 mg/m2 daily dose (Experimental): Pediatric dose.
  Interventions: Drug: LDE225
- LDE225 800 mg/m2 daily dose (Experimental): Adult dose
  Interventions: Drug: LDE225

INTERVENTIONS:
Drug: LDE225 — LDE225/sonidegib capsules were supplied to the Investigators at dose strengths of 50 mg, 100 mg, 200 mg, and 250 mg.
  Other Names: sonidegib

SUMMARY:
Phase I dose-escalation study to characterize the safety, tolerability, pharmacokinetics and pharmacodynamics of LDE225 given orally on a daily dosing schedule in children with recurrent or refractory medulloblastoma, or other tumors potentially dependent on Hedgehog signaling pathway.

Phase II study is to assess preliminary efficacy in both adult and pediatric patients with recurrent or refractory MB.

ELIGIBILITY:
Inclusion Criteria:

* Phase I - Patients aged ≥12 months and <18 years, Phase II - Patients ≥12 months
* Phase I - Histologically confirmed diagnosis of medulloblastoma, rhabdomyosarcoma, neuroblastoma, hepatoblastoma, high grade glioma, or osteosarcoma, that has progressed despite treatment with standard therapies, or for which no standard treatments are available (patients with brainstem gliomas are excluded). Phase II - Histologically confirmed diagnosis of recurrent or relapsed medulloblastoma with at least one measurable lesion.
* Performance Status: Karnofsky ≥60% for patients >10 yrs, Lansky ≥50 for patients less than or equal to 10 yrs
* Protocol-defined renal , liver and bone marrow function
* Negative pregnancy test before starting study treatment. If of child bearing potential must use 'highly effective' methods of contraception.
* All patients must consent to provide a tumor sample

Exclusion Criteria:

* Systemic anti-cancer treatment within 2 weeks prior to first dose (6 weeks for nitrosourea, mitomycin and monoclonal antibodies).
* Focal radiotherapy within 4 weeks prior to first dose, or full spinal radiotherapy within 3 months of first dose.
* Unresolved toxicity greater than CTCAE grade 1 from previous anti-cancer therapy or radiotherapy (excluding neurotoxicity, alopecia, ototoxicity, lymphopenia or other specifications in the eligibility criteria for this study), or incomplete recovery from previous surgery, unless agreed by Novartis and the Principal Investigator (PI) and documented.
* Major surgery, serious illness or traumatic injury within 2 weeks of starting study therapy. Patients anticipated to require major surgery within the first 2 cycles of treatment.
* Patients requiring a nasogastric tube for drug administration (G-tubes are permitted)
* Impaired cardiac function
* Pregnant or breast-feeding females
* Impairment of gastrointestinal (GI) function or GI disease

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 12 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 76 (Actual)
Dates: Start 2011-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (13):
- United States (4):
  - Children's Healthcare of Atlanta Childern Hosp - ATL, Atlanta, Georgia
  - Sidney Kimmel Comprehensive Cancer Center/Johns Hopkins Med. John Hopkins, Baltimore, Maryland
  - Dana Farber Cancer Institute DFCI (3), Boston, Massachusetts
  - Seattle Children's Hospital CPKC412A2114, Seattle, Washington
- Novartis Investigative Site, Parkville, Victoria, Australia
- Novartis Investigative Site, Toronto, Ontario, Canada
- France (2):
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Villejuif
- Italy (3):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Roma, RM
- United Kingdom (2):
  - Novartis Investigative Site, Sutton, Surrey
  - Novartis Investigative Site, Newcastle upon Tyne

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 14 centers in 6 countries.
Pre-assignment Details: A total of 76 participants: 60 pediatric and 16 adult participants were enrolled in this study, of which 59 pediatric participants received sonidegib during the dose-escalation and expansion part (Phase I); 17 participants (1 child and 16 adults) received sonidegib in the Phase II.
Groups:
- Pediatric Participants, LDE225 233 mg/m^2: Pediatric Participants received LDE225 233 mg/m^2 once daily through oral route.
- Pediatric Participants, LDE225 372 mg/m^2: Pediatric Participants received LDE225 372 mg/m^2 once daily through oral route.
- Pediatric Participants, LDE225 425 mg/m^2: Pediatric Participants received LDE225 425 mg/m^2 once daily through oral route.
- Pediatric Participants, LDE225 680 mg/m^2: Pediatric Participants received LDE225 680 mg/m^2 once daily through oral route. The Phase I , Phase II patients are pooled and summarized by dose levels. One pediatric patient enrolled in the Phase II portion at the 680 mg/m2 dose was pooled with 21 pediatric patients enrolled in Phase I at the same dose
- Adult Participants, LDE225 800 mg: Adult Participants were treated with LDE225 800 mg capsule once daily.
Period: Phase I
Arm/Group | Pediatric Participants, LDE225 233 mg/m^2 | Pediatric Participants, LDE225 372 mg/m^2 | Pediatric Participants, LDE225 425 mg/m^2 | Pediatric Participants, LDE225 680 mg/m^2 | Adult Participants, LDE225 800 mg
Started | 11 | 16 | 11 | 21 | 0 (None of participants were enrolled to this treatment in this period.)
Completed | 3 | 7 | 7 | 10 | 0
Not Completed | 8 | 9 | 4 | 11 | 0
Not completed — Protocol Violation | 0 | 3 | 1 | 1 | 0
Not completed — Adverse Event | 2 | 2 | 1 | 7 | 0
Not completed — Administrative problems | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0
Not completed — Disease progression | 5 | 4 | 1 | 3 | 0
Period: Phase II
Arm/Group | Pediatric Participants, LDE225 233 mg/m^2 | Pediatric Participants, LDE225 372 mg/m^2 | Pediatric Participants, LDE225 425 mg/m^2 | Pediatric Participants, LDE225 680 mg/m^2 | Adult Participants, LDE225 800 mg
Started | 0 (None of participants were enrolled to this treatment in this period.) | 0 (None of participants were enrolled to this treatment in this period.) | 0 (None of participants were enrolled to this treatment in this period.) | 1 (None of participants were enrolled to this treatment in this period.) | 16 (Additional participants were enrolled to this treatment in this period.)
Completed | 0 | 0 | 0 | 0 | 5
Not Completed | 0 | 0 | 0 | 1 | 11
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2
Not completed — Disease progression | 0 | 0 | 0 | 1 | 8

BASELINE CHARACTERISTICS:
Population: The analysis was performed in full analysis set population, defined as all the participants who received at least one dose of sonidegib.
Groups:
- Pediatric Participants, LDE225 680 mg/m^2: Pediatric Participants received LDE225 680 mg/m^2 once daily through oral route.
- Total: Total of all reporting groups
Arm/Group | Pediatric Participants, LDE225 233 mg/m^2 | Pediatric Participants, LDE225 372 mg/m^2 | Pediatric Participants, LDE225 425 mg/m^2 | Pediatric Participants, LDE225 680 mg/m^2 | Adult Participants, LDE225 800 mg | Total
Number analyzed (Participants) | 11 | 16 | 11 | 22 | 16 | 76
Age, Customized [Number; unit: participants]
  ≤ 10 years | 4 | 3 | 5 | 11 | 0 | 23
  >10 years to 17 years | 7 | 13 | 6 | 11 | 0 | 37
  18-65 years | 0 | 0 | 0 | 0 | 16 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 3 | 10 | 7 | 30
  Male | 7 | 10 | 8 | 12 | 9 | 46

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLT) in Phase I
Description: DLT was defined as an adverse event (AE) or abnormal laboratory value assessed as unrelated to disease, disease progression, intercurrent illness, or concomitant medications. DLT included any grade 3 or 4 clinically-evident toxicity, Hematology: ≥ CTCAE grade 3 neutropenia (ANC <1.0x10^9/L); ≥ CTCAE grade 3 thrombocytopenia (platelets <50x10^9/L); ≥ CTCAE grade 3 anemia (Hgb <80 g/L); Febrile neutropenia (ANC <1x10^9/L, fever ‡ 38.5°C), Renal: ≥ CTCAE grade 3 serum creatinine (>3xULN), Hepatic: ≥ CTCAE grade 3 total bilirubin (>3xULN); ≥ 10xULN ALT elevation; grade 2 total bilirubin (>1.5ULN) together with ≥ grade 3 ALT elevation (>5xULN), Cardiac: ≥ CTCAE grade 3, Other AEs: ≥ CTCAE grade 3 vomiting or nausea despite optimal antiemetic therapy, diarrhea despite optimal antidiarrheal treatment.
Time Frame: Baseline, End of dose escalation part (Day 42)
Population: The analysis was performed in full analysis set (FAS), defined as all the participants who received at least one dose of sonidegib.
Measure: Number; unit: participants
Arm/Group | Pediatric Participants, LDE225 233 mg/m^2 | Pediatric Participants, LDE225 372 mg/m^2 | Pediatric Participants, LDE225 425 mg/m^2 | Pediatric Participants, LDE225 680 mg/m^2
Number analyzed (Participants) | 11 | 16 | 11 | 22
participants | 0 | 1 | 0 | 0

2. Primary Outcome: Maximum Tolerated Dose (MTD) of Sonidegib for Prolonged Use
Description: MTD was defined as highest dose level for which no more than 1 participant in a dose cohort experienced dose-limiting toxicity (DLT), based on Bayesian logistic regression model (BLRM) employing the escalation with overdose control (EWOC) principle. DLT was defined as an adverse event (AE) or abnormal laboratory value assessed as unrelated to disease, disease progression, intercurrent illness, or concomitant medications.k
Time Frame: Baseline, End of dose escalation part (Day 42)
Population: The MTD for the pediatric population was not established in this study. MTD was not achieved since 1 or no DLT was observed. The recommended phase II dose was established based on the safety, pharmacokinetics, and clinical responses observed.
Measure: Number; unit: mg/m^2
Groups:
- All Participants: All participants received LDE225 233, 372, 425, 680, 800 mg/m^2 once daily through oral route until disease progression, unacceptable toxicity, or consent withdrawal.
Arm/Group | All Participants
Number analyzed (Participants) | 60
mg/m^2 | 680

3. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Treatment Related AEs and Death During the Study
Description: An AE was defined as any unfavorable and unintended sign, symptom, or disease temporally associated with the use of study drug, whether or not related to study drug. A SAE was defined as an event which was fatal or life threatening, required or prolonged hospitalization, was significantly or permanently disabling or incapacitating, constituted a congenital anomaly or a birth defect, or encompassed any other clinically significant event that could jeopardize the participant or require medical or surgical intervention to prevent one of the aforementioned outcomes. Treatment related AEs were defined as AEs that were suspected to be related to study treatment as per investigator. On-treatment deaths were deaths which occurred up to 30 days after last date of study treatment.
Time Frame: Baseline (start of study treatment) up to End of treatment (Within 14 days of last dose)
Population: The analysis was performed in safety set (SS), defined as all the participants who received at least 1 dose of sonidegib.
Measure: Number; unit: participants
Arm/Group | Pediatric Participants, LDE225 233 mg/m^2 | Pediatric Participants, LDE225 372 mg/m^2 | Pediatric Participants, LDE225 425 mg/m^2 | Pediatric Participants, LDE225 680 mg/m^2 | Adult Participants, LDE225 800 mg
Number analyzed (Participants) | 11 | 16 | 11 | 22 | 16
participants
  AEs | 11 | 16 | 11 | 22 | 16
  AEs suspected to be drug related | 8 | 13 | 9 | 14 | 13
  AEs leading to discontinuation | 1 | 1 | 1 | 1 | 3
  On-treatment deaths | 2 | 2 | 1 | 8 | 2
  SAEs | 5 | 8 | 4 | 14 | 5

4. Secondary Outcome: Area Under the Drug Concentration Time Curve From Time Zero to 24 Hours After Dosing (AUC0-24h) of Sonidegib in Phase I
Description: AUC(0-24h) was defined as the area under the drug concentration time curve calculated using linear trapezoidal summation from time zero to 24 hours after dosing.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 7 hours (± 15 min) post-dose at Day 1 and Day 22 of Cycle 1
Population: The analysis was performed in pharmacokinetic analysis set (PAS), defined as all the participants who received at least one (full or partial) dose of sonidegib and provided at least one evaluable pharmacokinetic (PK) blood sample. The 'n' signifies those participants evaluable for this measure at specified time points for each group, respectively.
Measure: Mean (Standard Deviation); unit: nanograms*hours/millilitres (ng*hr/mL)
Arm/Group | Pediatric Participants, LDE225 233 mg/m^2 | Pediatric Participants, LDE225 372 mg/m^2 | Pediatric Participants, LDE225 425 mg/m^2 | Pediatric Participants, LDE225 680 mg/m^2
Number analyzed (Participants) | 11 | 16 | 11 | 22
nanograms*hours/millilitres (ng*hr/mL)
  Cycle 1/Day 1 (n=11, 15, 11, 19) | 1981.56 (736.928) | 2194.29 (1592.396) | 5309.44 (3247.088) | 5117.61 (2658.133)
  Cycle 1/Day 22 (n=9, 14, 9, 15) | 10589.53 (4163.192) | 15431.43 (10433.35) | 17753.32 (11551.57) | 32622.67 (11670.63)

5. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Sonidegib in Phase I
Description: Tmax was defined as the time required to reach maximum observed plasma concentration. Tmax was directly determined from the raw plasma concentration time data.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 7 hours (± 15 min) post-dose at Day 1 and Day 22 of Cycle 1
Population: The analysis was performed in PAS population. The 'n' signifies those participants evaluable for this measure at specified time points for each group, respectively.
Measure: Median (Full Range); unit: hours
Arm/Group | Pediatric Participants, LDE225 233 mg/m^2 | Pediatric Participants, LDE225 372 mg/m^2 | Pediatric Participants, LDE225 425 mg/m^2 | Pediatric Participants, LDE225 680 mg/m^2
Number analyzed (Participants) | 11 | 16 | 11 | 22
hours
  Cycle 1/Day 1 (n=11, 15, 10, 17) | 3.98 [1.07 to 6.75] | 2.03 [1 to 7] | 2.92 [0.5 to 7] | 2.08 [1 to 4.08]
  Cycle 1/Day 22 (n=9, 12, 9, 15) | 1.98 [1 to 7] | 2.06 [0.95 to 4.25] | 2 [0.67 to 7] | 2 [0 to 7.05]

6. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Sonidegib in Phase I
Description: Maximum observed plasma concentration following drug administration was calculated from the raw plasma concentration time data.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 7 hours (± 15 min) post-dose at Day 1 and Day 22 of Cycle 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: nanograms/millitres(ng/mL)
Arm/Group | Pediatric Participants, LDE225 233 mg/m^2 | Pediatric Participants, LDE225 372 mg/m^2 | Pediatric Participants, LDE225 425 mg/m^2 | Pediatric Participants, LDE225 680 mg/m^2
Number analyzed (Participants) | 11 | 16 | 11 | 22
nanograms/millitres(ng/mL)
  Cycle 1/Day 1 (n=11, 15, 10, 17) | 191.18 (82.464) | 246.39 (211.034) | 642.5 (486.709) | 618.88 (403.466)
  Cycle 1/Day 22 (n=9, 12, 9, 15) | 769.22 (496.021) | 944.17 (553.395) | 1122 (736.862) | 1930 (677.949)

7. Secondary Outcome: Percentage of Pediatric Participants With Objective Response Rate (ORR) by Hedgehog (Hh) Signaling Pathway Status
Description: ORR was determined in the participants with mutations on Hh gene (Hh positive) and the participants without mutations on Hh gene (Hh negative).
Time Frame: Baseline, Day 28 of Cycle 2, End of treatment (Within 14 days of last dose)
Population: 60 patients with known (Hedgehog) Hh pathway activation status were analyzed, 10 patients, including all 5 patients with an objective response (3 with pediatric) , were Hh-positive (+). No Hh-negative patient had an objective response.
Measure: Number; unit: % pediatric Hh + responders
Groups:
- Pediatric Participants: All the pediatric Participants were treated with LDE225 dose determined in the Phase I (233, 372, 425 and 680 mg/m^2).
Arm/Group | Pediatric Participants
Number analyzed (Participants) | 3
% pediatric Hh + responders | 66.7

8. Secondary Outcome: Duration of Response by Treatment
Description: Duration of overall response (complete response (CR) or partial response (PR)) was calculated for those participants whose best overall response was CR or PR. The start date was the date of the first documented tumor response (CR or PR) and the end date was the date of the event defined as the first documented progression or death due to underlying cancer or after the same treatment line. If a participant did not have a progression or death, the duration of response was censored at the date of last adequate tumor assessment in that treatment line.
Time Frame: Baseline, Day 28 of Cycle 2, End of treatment (Within 14 days of last dose)
Population: The analysis was performed in FAS population. Here "Number of participants analysed" signifies treatment responders for the specified reporting group.
Measure: Median (Full Range); unit: months
Arm/Group | Pediatric Participants, LDE225 233 mg/m^2 | Pediatric Participants, LDE225 372 mg/m^2 | Pediatric Participants, LDE225 425 mg/m^2 | Pediatric Participants, LDE225 680 mg/m^2 | Adult Participants, LDE225 800 mg
Number analyzed (Participants) | 0 | 1 | 1 | 0 | 3
months |  | 7 [7 to 7] | 8.1 [8.1 to 8.1] |  | 4.86 [4.6 to 8.7]

9. Primary Outcome: Percentage of Participants With Objective Response Rate (ORR) by Treatment
Description: The tumor response to the sonidegib treatment was measured by ORR. The ORR was defined as the percentage of participants with partial response or complete response as their best overall response. Participants with stable disease, progressive disease tumor assessment were considered as non-responders. Response evaluation criteria was gadolinium chelate-enhanced brain tumor magnetic resonance imaging (Gd-MRI) for Medulloblastoma and central nervous system (CNS) tumors and response evaluation criteria in solid tumors (RECIST) version 1.0 for non-CNS tumors assessed by MRI. Complete Response (CR), Progressive Disease (PD) and Incomplete Response/Stable Disease (SD) were defined as disappearance of all non-target lesions, unequivocal progression of existing non-target lesions and Neither CR nor PD, respectively.
Time Frame: Baseline, Day 28 of Cycle 2, End of treatment (Within 14 days of last dose)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Groups:
- Adult Participants: All adult Participants were treated with sonidegib 800 mg once daily in phase II portion of the study. Pediatric patients were also enrolled in phase II portion of the study at the recommended phase II pediatric dose - 680 mg/m^2
Arm/Group | Pediatric Participants | Adult Participants
Number analyzed (Participants) | 60 | 16
Percentage of participants
  Complete response | 3.3 | 12.5
  Partial response | 0 | 6.3
  Stable disease | 8.3 | 37.5
  Progressive disease | 76.7 | 37.5
  Objective response rate | 3.3 | 18.8

ADVERSE EVENTS:
Time Frame: Adverse Events are collected from First Participant First Visit (FPFV) until Last Participant Last Visit (LPLV), Week 73. All Adverse events are reported in this record from First Participant First Treatment until LPLV, Week 73.
Arm/Group | Pediatric Participants, LDE225 233 mg/m^2 | Pediatric Participants, LDE225 372 mg/m^2 | Pediatric Participants, LDE225 425 mg/m^2 | Pediatric Participants, LDE225 680 mg/m^2 | Adult Participants, LDE225 800 mg
Serious Adverse Events (participants affected / at risk) | 5/11 | 8/16 | 4/11 | 14/22 | 5/16
Other Adverse Events (participants affected / at risk) | 11/11 | 16/16 | 11/11 | 21/22 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pediatric Participants, LDE225 233 mg/m^2 (N=11) | Pediatric Participants, LDE225 372 mg/m^2 (N=16) | Pediatric Participants, LDE225 425 mg/m^2 (N=11) | Pediatric Participants, LDE225 680 mg/m^2 (N=22) | Adult Participants, LDE225 800 mg (N=16)
Vision Blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 4 | 0
Chest Pain (General disorders) | 0 | 1 | 0 | 0 | 0
General Physical Health Deterioration (General disorders) | 1 | 2 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 2 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Mucosal Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Wound Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Procedural Complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 0 | 1
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood Creatine Phosphokinase Increased (Investigations) | 0 | 0 | 0 | 0 | 2
Myoglobin Blood Increased (Investigations) | 0 | 0 | 0 | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Altered State Of Consciousness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Coma (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 0 | 3 | 0
Depressed Level Of Consciousness (Nervous system disorders) | 0 | 0 | 0 | 2 | 0
Dysaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Dystonia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 1 | 4 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Intracranial Pressure Increased (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Neurological Decompensation (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Quadriparesis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
VIIth Nerve Paralysis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Confusional State (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0
Disorientation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Suicidal Ideation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Urinary Incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Venous Insufficiency (Vascular disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pediatric Participants, LDE225 233 mg/m^2 (N=11) | Pediatric Participants, LDE225 372 mg/m^2 (N=16) | Pediatric Participants, LDE225 425 mg/m^2 (N=11) | Pediatric Participants, LDE225 680 mg/m^2 (N=22) | Adult Participants, LDE225 800 mg (N=16)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 4 | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 2 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Left Ventricular Hypertrophy (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Sinus Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cerumen Impaction (Ear and labyrinth disorders) | 2 | 0 | 0 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Ear Canal Stenosis (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Ear Pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Cushingoid (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
Blindness Unilateral (Eye disorders) | 1 | 0 | 0 | 0 | 0
Conjunctivitis Allergic (Eye disorders) | 0 | 0 | 1 | 0 | 0
Diplopia (Eye disorders) | 0 | 1 | 0 | 0 | 0
Dry Eye (Eye disorders) | 0 | 0 | 1 | 1 | 0
Eye Irritation (Eye disorders) | 0 | 0 | 1 | 0 | 0
Eyelid Ptosis (Eye disorders) | 0 | 1 | 0 | 0 | 0
Lacrimation Increased (Eye disorders) | 0 | 1 | 0 | 1 | 0
Ocular Hyperaemia (Eye disorders) | 0 | 1 | 0 | 0 | 0
Strabismus (Eye disorders) | 0 | 0 | 1 | 1 | 0
Vision Blurred (Eye disorders) | 0 | 1 | 2 | 1 | 0
Visual Acuity Reduced (Eye disorders) | 0 | 0 | 1 | 0 | 0
Visual Impairment (Eye disorders) | 1 | 0 | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 3 | 2 | 5 | 1
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Anal Pruritus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 6 | 4 | 3 | 2
Dental Caries (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 5 | 2 | 1 | 4
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 1
Faecal Incontinence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Faeces Hard (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastrointestinal Pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gingival Pain (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Mouth Ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 5 | 4 | 3 | 8 | 4
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Oral Dysaesthesia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Oral Pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 3
Tooth Disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 5 | 9 | 7 | 15 | 2
Asthenia (General disorders) | 2 | 4 | 1 | 1 | 3
Chest Pain (General disorders) | 0 | 2 | 0 | 1 | 0
Chills (General disorders) | 1 | 0 | 0 | 0 | 0
Face Oedema (General disorders) | 0 | 1 | 0 | 0 | 0
Facial Pain (General disorders) | 0 | 1 | 0 | 0 | 1
Fatigue (General disorders) | 5 | 7 | 3 | 6 | 1
Gait Disturbance (General disorders) | 1 | 1 | 1 | 1 | 2
General Physical Health Deterioration (General disorders) | 0 | 0 | 0 | 0 | 1
Influenza Like Illness (General disorders) | 0 | 0 | 0 | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 1 | 0 | 0
Oedema Peripheral (General disorders) | 0 | 2 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1 | 1 | 0
Performance Status Decreased (General disorders) | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 3 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0
Catheter Site Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 1 | 0 | 1 | 1
Ear Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Skin Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Tooth Abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 2
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 1 | 1 | 1
Vulvovaginal Mycotic Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Vascular Procedure Complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Activated Partial Thromboplastin Time Prolonged (Investigations) | 0 | 1 | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 2 | 0 | 2 | 4
Aspartate Aminotransferase Increased (Investigations) | 0 | 2 | 2 | 2 | 1
Blood Alkaline Phosphatase Increased (Investigations) | 1 | 1 | 1 | 0 | 0
Blood Bilirubin Increased (Investigations) | 0 | 0 | 0 | 1 | 1
Blood Creatine Phosphokinase Increased (Investigations) | 1 | 1 | 2 | 6 | 8
Blood Creatinine Increased (Investigations) | 0 | 0 | 1 | 1 | 0
Blood Fibrinogen Decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood Lactate Dehydrogenase Increased (Investigations) | 2 | 0 | 0 | 0 | 0
Blood Magnesium Decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood Urea Increased (Investigations) | 1 | 0 | 0 | 0 | 0
Cardiac Murmur (Investigations) | 0 | 1 | 0 | 0 | 0
Haemoglobin Decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Lymphocyte Count Decreased (Investigations) | 2 | 1 | 3 | 3 | 1
Neutrophil Count Decreased (Investigations) | 0 | 2 | 2 | 2 | 0
Platelet Count Decreased (Investigations) | 0 | 2 | 1 | 0 | 0
Weight Decreased (Investigations) | 1 | 2 | 0 | 2 | 3
White Blood Cell Count Decreased (Investigations) | 2 | 2 | 3 | 3 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 1 | 3 | 4 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyperphagia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 3 | 1 | 3 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 0
Vitamin D Deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 3 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0 | 0 | 1
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Epiphyseal Disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 | 4 | 5 | 2 | 4
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 0
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 4 | 5 | 5
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 2 | 1 | 2
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 2 | 6 | 4 | 0 | 0
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0 | 1
Posture Abnormal (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Sensation Of Heaviness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Temporomandibular Joint Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 2 | 0 | 1 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Ataxia (Nervous system disorders) | 2 | 2 | 2 | 4 | 0
Balance Disorder (Nervous system disorders) | 1 | 0 | 1 | 0 | 1
Brain Oedema (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Cerebellar Syndrome (Nervous system disorders) | 0 | 1 | 0 | 1 | 1
Coma (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 2 | 2 | 1
Coordination Abnormal (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Depressed Level Of Consciousness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 0 | 0
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Facial Nerve Disorder (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Facial Paresis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 6 | 7 | 4 | 9 | 2
Hemiparesis (Nervous system disorders) | 0 | 0 | 1 | 3 | 0
Hemiplegia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 2 | 0 | 0 | 0
III rd Nerve Paresis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Intracranial Pressure Increased (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 3 | 0 | 0
Meningism (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Neurological Decompensation (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Neuropathy Peripheral (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 2
Paraparesis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Peroneal Nerve Palsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Pyramidal Tract Syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 3 | 1 | 1 | 0
Speech Disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
VII th Nerve Paralysis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
VI th Nerve Disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 2 | 1 | 1 | 0
Bruxism (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Confusional State (Psychiatric disorders) | 1 | 2 | 1 | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Euphoric Mood (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 2 | 1 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0
Mood Altered (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Paranoia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0
Micturition Disorder (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Micturition Urgency (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Neurogenic Bladder (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 1 | 1 | 1
Polyuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urinary Incontinence (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 1
Urinary Retention (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0
Urinary Tract Disorder (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Penile Pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Vaginal Discharge (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 5 | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 3
Laryngeal Inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 3 | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Fungating Wound (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Madarosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 0 | 0
Nail Disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Pain Of Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 3 | 1 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash Papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Solar Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 2 | 0 | 1 | 1
Pallor (Vascular disorders) | 0 | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
The Phase I and Phase II patients are pooled and summarized by dose levels. One pediatric patient enrolled in the Phase II portion at the 680 mg/m2 dose was pooled with 21 pediatric patients enrolled in Phase I at the same dose

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single--site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.